CLINICAL TRIAL: NCT05440305
Title: Castleman Disease - Diagnosis and Surgery
Brief Title: Unicentric Form of Castleman Disease - Surgery Therapy Benefit
Status: Completed | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jiri Molacek, Principal investigator, Charles University, Czech Republic
Other Study IDs: 750923
Record Dates: First submitted 2022-05-11; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Castleman Disease; Unicentric Castleman Disease; Surgery
Keywords: Unicentric form of Castleman disease; Surgical resection
MeSH Terms: conditions — Castleman Disease; Angiolymphoid Hyperplasia with Eosinophilia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery type/exstirpation/debulking — Evaluation of benefit according to surgery

SUMMARY:
Observation study on patients with unicentric form of Castleman disease, evaluation of surgical treatment benefit. Observation of surgical treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* patient with unicentric form of Castleman disease
* underwent surgery resection

Exclusion Criteria:

* multilocalised Castleman disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group of patients with unicentric form of Castleman disease
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
5 year survival | each 6 months checkup, up to 150 weeks, from date of randomization until the date of first documented progression
  surgery treatment success
recurence rate | each 6 months checkup, up to 150 weeks, from date of randomization until the date of first documented progression
  surgery treatment success

IPD SHARING:
Plan to Share IPD: No